CLINICAL TRIAL: NCT03388476
Title: Endtidal Carbon Dioxide for Earlier Detection of Pulmonary Hypertension in Patients With Suspicion of Pulmonary Hypertension
Brief Title: Endtidal Carbon Dioxide for Earlier Detection of Pulmonary Hypertension
Acronym: EARLIER
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Sophie Herbst, Study Chair: Ghofrani H. Ardeschir, Prof. Dr. University of Giessen, University of Giessen
Other Study IDs: AZ 156/17; DRKS00013589 (Registry Identifier: DRKS); AZ 156/17 (Other: Ethik-Kommission Giessen)
Record Dates: First submitted 2017-12-22; First posted 2018-01-03 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Hypertension, Pulmonary; Hypertension;Pulmonary;Primary; Chronic Thromboembolic Pulmonary Hypertension; Vascular Diseases; Lung Diseases
Keywords: pulmonary hypertension; endtidal co2; endtidal carbon dioxide; pulmonary arterial hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Familial Primary Pulmonary Hypertension; Vascular Diseases; Lung Diseases; Pulmonary Arterial Hypertension | interventions — Capnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspicion of pulmonary hypertension: At Patients with suspicion of pulmonary hypertension, which get a right heart catheterization, in the context of the study the exhaled air, precious the endtidal carbon dioxide (CO2), before or after the right heart catheterization will be measured through capnography.
  Interventions: Diagnostic Test: Capnography

INTERVENTIONS:
Diagnostic Test: Capnography — Measuring of the exhaled air, especially endtidal co2, through capnography.

SUMMARY:
Measurement of the endtidal carbon dioxide by capnography to exclude or to ensure the diagnosis pulmonary hypertension. The aim of the study is to obtain an endtidal carbon dioxide cut-off value for the diagnostic algorithm for pulmonary hypertension as an easily measurable and cheap diagnostic tool in patients with suspicion of pulmonary hypertension.

DETAILED DESCRIPTION:
The disease pulmonary hypertension is due to a remodeling of the lung vessels which results in a change of the exhaled air. This change is measurable with a so called capnograph. The investigators want to measure the breath from patients with and without pulmonary hypertension to detect a cut-off value for the diagnosis pulmonary hypertension.

Patients which have the probably diagnosis pulmonary hypertension and are older than 18 years are investigated. This patients will get an right heart catheterization and a measurement from their exhaled air.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years, suspicion of pulmonary hypertension, planned or accomplished right heart catheterization

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of a tertiary referral center retro- and prospective part of the study.
  Afterwards in a next prospective study part patients in ambulant setting.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Measurement PetCO2 | At baseline
  Measurement PetCO2 by capnography at rest after or before a right heart catheterization, comparison of the parameter between patients with and without

SECONDARY OUTCOMES:
Establishing a cut-off | At baseline
  Establishing a cut-off for the non-invasive diagnosing of pulmonary hypertension, which differs between patients with and without pulmonary hypertension and save patients without the disease before a dispensable invasive right heart catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Henning Gall, MD, PhD, Principal Investigator — University Clinic Giessen and Marburg - Campus Giessen; Werner Seeger, Prof., Study Director — University Clinic Giessen and Marburg; Ardeschir Ghofrani, Prof., Study Director — University Clinic Giessen and Marburg
Locations (1):
- University Clinic Giessen and Marburg, Giessen, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hemnes AR, Pugh ME, Newman AL, Robbins IM, Tolle J, Austin ED, Newman JH. End tidal CO(2) tension: pulmonary arterial hypertension vs pulmonary venous hypertension and response to treatment. Chest. 2011 Nov;140(5):1267-1273. doi: 10.1378/chest.11-0155. Epub 2011 May 26. PMID 21622547